CLINICAL TRIAL: NCT07126730
Title: Investigating the Effects of the EXOPULSE Mollii Suit on Spasticity and Functionality in Patients With Multiple Sclerosis
Brief Title: Effects of EXOPULSE Mollii Suit on Spasticity and Functionality in Multiple Sclerosis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Muhammed KILINÇ, Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FTREK25/78
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: spasticity; delete
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXOPULSE Mollii + Exercise (Experimental): During the 60-minute EXOPULSE Mollii stimulation session, patients will also perform a guided exercise program.
  Interventions: Device: EXOPULSE Mollii Suit + Exercise
- EXOPULSE Mollii (Active Comparator): For 60 minutes, patients will only receive stimulation while wearing the EXOPULSE Mollii suit.
  Interventions: Device: EXOPULSE Mollii Suit

INTERVENTIONS:
Device: EXOPULSE Mollii Suit + Exercise — First, spasticity will be evaluated using the Modified Ashworth Scale (MAS). Based on this evaluation, the stimulation intensity for each muscle group will be determined and recorded in the system. Once patients put on the EXOPULSE Mollii Suit and the stimulation begins, they will undergo a personalized exercise program including strengthening, balance, and gait training with scheduled rest intervals. All MS patients will undergo treatment three days per week (with at least one day between sessions) for one hour per day over four weeks.
  Arms: EXOPULSE Mollii + Exercise
Device: EXOPULSE Mollii Suit — First, spasticity will be evaluated using the Modified Ashworth Scale (MAS). Based on this evaluation, the stimulation intensity for each muscle group will be determined and recorded in the system. Patients will wear the suit and receive stimulation while resting for 60 minutes. All MS patients will undergo treatment three days per week (with at least one day between sessions) for one hour per day over four weeks.
  Arms: EXOPULSE Mollii

SUMMARY:
Spasticity affects >80% of MS patients, with 35-54% experiencing moderate-to-severe symptoms, impairing mobility and sleep. Electrical stimulation parameters (e.g., high vs. low frequency) for spasticity management remain debated. The EXOPULSE Mollii Suit uses non-invasive, low-frequency stimulation to induce reciprocal inhibition and modulate spinal interneuron activity, potentially reducing spasticity. This study aims to compare EXOPULSE Mollii + exercise vs. EXOPULSE Mollii alone in improving spasticity and function in MS.

DETAILED DESCRIPTION:
Spasticity is one of the most common symptoms in multiple sclerosis (MS) patients. Large-scale surveys indicate that over 80% of MS patients experience spasticity during their disease course, with 35-54% reporting moderate to severe spasticity. Spasticity, particularly in the lower extremities, is associated with stiffness, spasms, and pain and negatively affects walking, stair climbing, and sleep. While electrical stimulation is a potential treatment for spasticity, optimal stimulation parameters remain unclear. The most commonly used protocol involves high-frequency stimulation (~100 Hz), though some studies suggest low-frequency stimulation may also be effective.

The EXOPULSE Mollii suit (EXONEURAL NETWORK AB, Danderyd, Sweden) is a non-invasive, self-administered electrical stimulation system with integrated electrodes. It is designed to reduce spasticity and improve motor function in neurological disorders. The method is based on reciprocal inhibition, where low-frequency, low-intensity stimulation of antagonist muscles activates Ia inhibitory interneurons, reducing spasticity in agonist muscles. Additional mechanisms may include neuroplastic changes in spinal or brain circuits, similar to transcutaneous electrical nerve stimulation (TENS). This study aims to compare the effects of EXOPULSE Mollii + exercise vs. EXOPULSE Mollii alone on spasticity and functionality in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MS by a neurologist according to McDonald criteria
* Age >18 years
* EDSS score ≤6.5 (able to walk independently without assistive devices)
* Presence of spasticity
* Mini Mental State Examination (MMSE) score ≥24

Exclusion Criteria:

* Received surgical intervention or botulinum toxin injection for spasticity within the last 6 months
* Presence of any neurological condition (other than MS) that may affect independent standing or walking
* Currently participating in another rehabilitation program
* Declined to participate or provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | 4 weeks
  Spasticity in patients will be assessed using the Modified Ashworth Scale (MAS). It grades spasticity based on the resistance exhibited by the muscle, using a scale of 0, 1, 1+, 2, 3, and 4.
Berg Balance Scale (BBS) | 4 weeks
  This 14-item scale is scored from 0 to 4 for each item. A score of 0 indicates inability to perform, while a score of 4 indicates normal performance. With a maximum total score of 56, higher scores indicate better balance ability.
OptoGait Gait Analysis System | 4 weeks
  During the test, the patient is asked to step onto the treadmill. They are then asked to adjust the treadmill speed to their preferred pace and walk for one minute. While walking on the treadmill, objective data related to their gait's time-distance characteristics is obtained. The evaluation takes five minutes.

SECONDARY OUTCOMES:
EDSS (Expanded Disability Status Scale) | 4 weeks
  The severity of the disease will be assessed using the Expanded Disability Status Scale (EDSS). This assessment is based on a clinician's interview and the patient's neurological status. A score of 0 represents normal neurological status, while a score of 10 indicates worsening MS. The next score after 0 is 1, and clinical deterioration is expressed in 0.5-point increments thereafter. The EDSS score is calculated using a rating scale of 0.0 to 4.0 for pyramidal, cerebellar, brainstem, sensory, visual, bowel-bladder, and mental functions. The rating is based on the patient's best performance without excessive effort. A score of 0-4 indicates independence; 6.0, unilateral support; 6.5, bilateral support; and 7.0 or higher, dependence.
Visual Analog Scale (VAS) for pain and fatigue | 4 weeks
  The Visual Analog Scale will be used to assess pain and fatigue. Patients will rate their pain and fatigue on a 10-cm line. "No pain-no fatigue" will be scored as 0 points, and "the worst pain imaginable-the worst fatigue" will be scored as 10 points.
Fatigue Severity Scale | 4 weeks
  The Fatigue Severity Scale (FSS) is a nine-item scale that measures the severity of fatigue and its impact on patients' activities and lifestyle. Each item is scored on a scale from 1 to 7. A score of 1 indicates strong disagreement with the statement, while a score of 7 indicates strong agreement. The lowest possible total score is 7, and the highest possible total score is 63. The higher the score, the greater the fatigue severity.
9-Hole Peg Test | 4 weeks
  A nine-hole peg test will be used to evaluate hand function. The time it takes individuals to insert and remove the nine pegs from the holes will be recorded. Participants will perform the test with both their dominant and non-dominant hands.
5 Times Sit to Stand Test | 4 weeks
  Functional strength of the lower extremities will be assessed using the Five Times Sit-to-Stand Test. For this test, a standard-sized chair with a backrest (43-45 cm) is used. The patient sits on the chair with their back against the backrest. Each repetition of sitting down and standing up is counted. The time it takes to complete five repetitions is recorded using a stopwatch.
Timed Up and Go (TUG) Test | 4 weeks
  The TUG test measures functional mobility skills and risk of falling. For this test, participants stand up from a chair, walk three meters, turn around, walk back, and sit down again. The time it takes to complete this task is used to determine functional mobility. Completing the task in ≤10 seconds indicates normal functional mobility. Completing it in <20 seconds indicates good mobility, meaning the individual can walk without assistive devices and go out alone. Completing it in <30 seconds indicates a mobility issue, meaning the individual needs to use assistive devices and cannot go out alone.
10 meter Walk Test | 4 weeks
  A 10-meter walking test will be performed to evaluate patients' walking ability. Participants will walk 10 meters, and their time will be recorded with a stopwatch. The average time will be calculated based on three repetitions. Walking speed (m/s) will be calculated by dividing the walking distance (10 meters) by the average time obtained. Walking speeds are categorized as follows: <0.4 m/s indicates ambulation within the home, 0.4-0.8 m/s indicates limited ambulation outside the home, and >0.8 m/s indicates ambulation outside the home.
12-Item Multiple Sclerosis Walking Scale | 4 weeks
  It assesses the patient's walking abilities over the past two weeks from their perspective. Each question is scored on a five-point scale. Patients are asked to rate themselves as follows: 1 = none; 2 = slight; 3 = moderate; 4 = severe; and 5 = very severe. A high score indicates difficulty walking.
Functional Independence Measure (FIM) | 4 weeks
  Activities daily living will be assessed using the Functional Independence Measure (FIM). The FIM consists of 18 items that cover self-care, sphincter control, mobility, movement, communication, and social interaction. Scores range from 18 to 126.
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | 4 weeks
  It is a measure created by adding 18 multiple sclerosis (MS)-specific items to the Short Form 36 (SF-36), which contains 36 questions related to overall quality of life. Patients receive two separate scores, one for physical health and one for mental health. Higher scores indicate better outcomes. The scale's subparameters include physical health, physical role limitations, emotional role limitations, pain, energy levels, perceived health, social functions, cognitive functions, sexual functions, and overall quality of life. Total mental and physical scores are calculated based on the different coefficients of each sub-parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed KILINÇ, Prof. Dr., Principal Investigator — Hacettepe University, Faculty of Physical Therapy and Rehabilitation

IPD SHARING:
Plan to Share IPD: No